CLINICAL TRIAL: NCT05051904
Title: Comparative Safety and Effectiveness of Warfarin, Dabigatran, and Rivaroxaban Among Japanese Patients With Non-valvular Atrial Fibrillation (NVAF) and Concomitant Coronary Artery Disease (CAD)
Brief Title: A Study Based on Japanese Medical Records That Looks at Bleeding Events in People With Atrial Fibrillation and Coronary Artery Disease Who Start Taking Either Dabigatran, Rivaroxaban, or Warfarin
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0308
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Warfarin: All eligible Japanese on-valvular atrial fibrillation (NVAF) patients with concomitant Coronary Artery Disease (CAD), who were prescribed with warfarin. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database, which covered all insurance types and a large population size.
  The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
- Dabigatran: All eligible Japanese on-valvular atrial fibrillation (NVAF) patients with concomitant Coronary Artery Disease (CAD), who were prescribed with dabigatran. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database, which covered all insurance types and a large population size.
  The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
- Rivaroxaban: All eligible Japanese on-valvular atrial fibrillation (NVAF) patients with concomitant Coronary Artery Disease (CAD), who were prescribed with rivaroxaban. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database, which covered all insurance types and a large population size.
  The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).

SUMMARY:
The study aims to evaluate the safety and effectiveness comparisons between warfarin, dabigatran, and rivaroxaban in routine clinical practice among Japanese non-valvular atrial fibrillation (NVAF) patients with concomitant coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age

* Has one year of look-back period prior to the index date (defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the study period)
* New users of warfarin, dabigatran, and rivaroxaban, defined as patients without historic use of any oral anticoagulants during the look-back period
* Has at least 1 diagnosis of NVAF during the look-back period prior to or on the index date
* Has at least 1 diagnosis of CAD during the look-back period prior to or on the index date

Exclusion Criteria:

* Diagnosed with end-stage renal disease, or undergo hemodialysis, or experience pregnancy during the study period
* Initiate warfarin, dabigatran, rivaroxaban due to valvular Atrial Fibrillation (AF), AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis, or rheumatic AF
* Underwent joint replacement procedures or diagnosed with venous thromboembolism during the look-back period prior to or on the index date
* Prescribed with more than 1 oral anticoagulation (OAC) on the index date
* Prescribed with more than 2 anti-platelet drugs per prescription (triple or quadruple anti-platelet use), or prescribed with any anti-platelet injection
* Patients with missing or ambiguous age or sex information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese patients with non-valvular atrial fibrillation and concomitant coronary artery disease
Sampling Method: Probability Sample
Enrollment: 39357 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim - International GmbH, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Chen Y, Gong X, Bao H. Real-world clinical outcomes of oral anticoagulants among Japanese patients with atrial fibrillation and concomitant coronary artery disease. Int J Cardiol Heart Vasc. 2023 Nov 2;49:101285. doi: 10.1016/j.ijcha.2023.101285. eCollection 2023 Dec. PMID 38020057
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Real world, non-interventional cohort study based on existing data from The Medical Data Vision Co. Ltd. (Tokyo, Japan). The study aimed to make safety and effectiveness comparisons between warfarin, dabigatran, and rivaroxaban in routine clinical practice among Japanese non-valvular atrial fibrillation (NVAF) patients with concomitant Coronary Artery Disease (CAD).
Pre-assignment Details: Every patient who fulfilled inclusion and exclusion criteria and agreed to participate in the study was selected until the required sample size was achieved.
Period: Overall Study
Arm/Group | Warfarin | Dabigatran | Rivaroxaban
Started | 12316 | 6712 | 20329
Crude | 12316 | 6712 | 20329
s-IPTW Adjusted (Balanced to account for potential confounding effects through an inverse probability of treatment weighting (IPTW) method) | 12231 | 6682 | 20422
Completed | 12316 | 6712 | 20329
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Eligible: patients fulfilling all inclusion criteria and no exclusion criteria (Crude)
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | Dabigatran | Rivaroxaban | Total
Number analyzed (Participants) | 12316 | 6712 | 20329 | 39357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.0 (10.2) | 71.8 (10.6) | 74.2 (10.6) | 74.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4448 | 1820 | 6411 | 12679
  Male | 7868 | 4892 | 13918 | 26678
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Measure Analysis Population Description: Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Fatal or Non-fatal Major Bleeding
Description: Incidence rate of fatal or non-fatal major bleeding per number of person-years, defined as any blood transfusion and/or any hospitalization with associated bleeding in all three patient groups. The incidence rate was reported as the number of events (counts the first event per patient) divided by the total number of person-years at risk during follow-up (1/(1000*person-years)).
Time Frame: From the cohort entry date (first prescription of the drug of interest) to the earliest occurrence of the event (discontinuation of drug of interest, switching to another Oral Anticoagulation, loss of follow-up, death, end of the study). Up to 9 years.
Population: Matched cohort of initiators of Dabigatran, Warfarin, Rivaroxaban using the inverse probability of treatment weighting (IPTW) method, identified from the Japan Medical Data Vision Co. Ltd. (MDV) database on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
Measure: Number (95% Confidence Interval); unit: Events per 1,000 person-years
Groups:
- Dabigatran - Matched With Warfarin Using the s-IPTW Method; Dabigatran - Matched With Rivaroxaban Using the s-IPTW Method: Matched cohort of patients with on-valvular atrial fibrillation (NVAF) with concomitant Coronary Artery Disease (CAD), who were prescribed with Dabigatran. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database. The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
- Warfarin - Matched With Dabigatran Using the s-IPTW Method; Warfarin - Matched With Rivaroxaban Using the s-IPTW Method: Matched cohort of patients with on-valvular atrial fibrillation (NVAF) with concomitant Coronary Artery Disease (CAD), who were prescribed with Warfarin. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database. The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
- Rivaroxaban - Matched With Warfarin Using the s-IPTW Method; Rivaroxaban - Matched With Dabigatran Using the s-IPTW Method: Matched cohort of patients with on-valvular atrial fibrillation (NVAF) with concomitant Coronary Artery Disease (CAD), who were prescribed with Rivaroxaban. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database. The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
Arm/Group | Dabigatran - Matched With Warfarin Using the s-IPTW Method | Warfarin - Matched With Dabigatran Using the s-IPTW Method | Rivaroxaban - Matched With Warfarin Using the s-IPTW Method | Warfarin - Matched With Rivaroxaban Using the s-IPTW Method | Dabigatran - Matched With Rivaroxaban Using the s-IPTW Method | Rivaroxaban - Matched With Dabigatran Using the s-IPTW Method
Number analyzed (Participants) | 6682 | 12231 | 20422 | 12231 | 6682 | 20422
Events per 1,000 person-years | 26 [22 to 31] | 52 [47 to 57] | 41 [38 to 44] | 52 [47 to 57] | 26 [22 to 31] | 41 [38 to 44]
Statistical Analysis 1: Comparison: Dabigatran - Matched With Warfarin Using the s-IPTW Method vs Warfarin - Matched With Dabigatran Using the s-IPTW Method; Test type: Other; p < 0.0001, Regression, Cox; Cox proportional hazard model with s-IPTW. 'Treatment' is the only Independent variable used to estimate the hazard ratios; Adjusted Hazard Ratio = 0.5, 95% CI 2-sided [0.402 to 0.622] — Hazard ratio <1 favors Dabigatran
Statistical Analysis 2: Comparison: Rivaroxaban - Matched With Warfarin Using the s-IPTW Method vs Warfarin - Matched With Rivaroxaban Using the s-IPTW Method; Test type: Other; p = 0.0004, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Adjusted Hazard Ratio = 0.784, 95% CI 2-sided [0.686 to 0.896] — Hazard ratio <1 favors Rivaroxaban
Statistical Analysis 3: Comparison: Dabigatran - Matched With Rivaroxaban Using the s-IPTW Method vs Rivaroxaban - Matched With Dabigatran Using the s-IPTW Method; Test type: Other; p < 0.0001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Adjusted Hazard Ratio = 0.637, 95% CI 2-sided [0.514 to 0.791] — Hazard ratio <1 favors Dabigatran

2. Secondary Outcome: Incidence Rate of Composite Outcome of Stroke/SE/MI/All-cause Mortality (Inpatient) /Major Bleeding/Major GI Bleeding/ICH
Description: Incidence rate of the Composite outcome of stroke/SE/MI/all-cause mortality (inpatient) /major bleeding/major GI bleeding (hospitalization due to gastrointestinal bleeding)/ICH (Intracraneal hemorrhage) per number of person-years. The incidence rate was reported as the number of events (counts the first event per patient) divided by the total number of person-years at risk during follow-up (1/(1000*person-years)). The propensity scores were estimated using the multivariable logistic regression model. Statistical analysis for comparisons: Dabigatran-Warfarin, and Rivaroxaban-Warfarin are presented as per protocol.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1,000 person-years
Groups:
- Rivaroxaban - Matched With Warfarin Using the s-IPTW Method: Rivaroxaban - matched with Warfarin using the s-IPTW method Matched cohort of patients with on-valvular atrial fibrillation (NVAF) with concomitant Coronary Artery Disease (CAD), who were prescribed with Rivaroxaban. From existing data from the Japan Medical Data Vision Co. Ltd. (MDV) database. The study period started on April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).
Arm/Group | Dabigatran - Matched With Warfarin Using the s-IPTW Method | Warfarin - Matched With Dabigatran Using the s-IPTW Method | Rivaroxaban - Matched With Warfarin Using the s-IPTW Method | Warfarin - Matched With Rivaroxaban Using the s-IPTW Method | Dabigatran - Matched With Rivaroxaban Using the s-IPTW Method | Rivaroxaban - Matched With Dabigatran Using the s-IPTW Method
Number analyzed (Participants) | 6682 | 12231 | 20422 | 12231 | 6682 | 20422
Events per 1,000 person-years | 213 [200 to 228] | 275 [264 to 288] | 228 [220 to 237] | 275 [264 to 288] | 213 [200 to 228] | 228 [220 to 237]
Statistical Analysis 1: Comparison: Dabigatran - Matched With Warfarin Using the s-IPTW Method vs Warfarin - Matched With Dabigatran Using the s-IPTW Method; Test type: Other; p < 0.0001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Adjusted Hazard Ratio = 0.78, 95% CI 2-sided [0.714 to 0.851] — Hazard ratio <1 favors Dabigatran
Statistical Analysis 2: Comparison: Rivaroxaban - Matched With Warfarin Using the s-IPTW Method vs Warfarin - Matched With Rivaroxaban Using the s-IPTW Method; Test type: Other; p < 0.0001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Adjusted Hazard Ratio = 0.827, 95% CI 2-sided [0.777 to 0.88] — Hazard ratio<1 favors Rivaroxaban

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data, safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Warfarin | Dabigatran | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a Non interventional study (NIS) based on existing data. Therefore, the study might be subject to potential residual confounding due to the absence of certain key data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05051904/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05051904/SAP_001.pdf